CLINICAL TRIAL: NCT06226675
Title: The Effect of Adding Lateral Femoral Cutaneous Nerve Block to PENG Block on Postoperative Opioid Consumption in Hip Surgery
Brief Title: 'The Effect of Adding LFCN Block to PENG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Keziban Bollucuoglu, Principal Investigator, Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020/15-14
Record Dates: First submitted 2024-01-04; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Pain, Postoperative; Pain, Acute; Nerve Block; Opioid Consumption
Keywords: lateral femoral cutaneous nerve block; PENG block; Pain management; Opioid consumption
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (No Intervention)
- Group PENG (Active Comparator)
  Interventions: Procedure: PENG Block
- Group PENG+LFCN (Active Comparator)
  Interventions: Procedure: PENG Block; Procedure: LFCN block

INTERVENTIONS:
Procedure: PENG Block — To apply local anesthetic under psoas tendon
  Arms: Group PENG; Group PENG+LFCN
Procedure: LFCN block — to apply local anesthetic around lateral femoral cutaneous nerve
  Arms: Group PENG+LFCN

SUMMARY:
The incidence of femoral neck fracture in Europe is 330/10000 per year. It is increasing every year due to the aging of the population. In patients 55 years and older, hip fracture-related mortality is estimated to be between 4% and 16% at one month and between 11% and 43% at one year after surgery. The reduced risk of postoperative complications associated with the use of regional anesthesia, shorter mobilization times, and reduced morphine consumption in hip fractures have been reported, and have been incorporated into postoperative pain control as part of multimodal strategies. PENG has been described for postoperative pain control for surgery on the hip joint or for the treatment of post-traumatic pain associated with proximal femur/femoral head fractures. Lateral femoral cutaneous nerve block is used in combination with other peripheral block methods to provide analgesia in the lateral thigh.

The investigators aimed to evaluate the effect of adding lateral femoral cutaneous nerve block to PENG block on pain scores and opioid consumption in femoral fracture procedures under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old,
* ASA I-II-III risk group
* patients undergoing hip fracture surgery under spinal anesthesia
* Patients whose informed consent was read and consent was obtained from them and their representatives.

Exclusion Criteria:

* Those who do not want to participate in the study,
* ASA IV-V patients
* Those with coagulation disorders
* Allergic to local anesthetics

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
postoperative opioid consumption | up to 24 hour after surgery
  total morphine requirement

SECONDARY OUTCOMES:
pain scores | up to 24 hour after surgery
  evaluating pain scores by Numeric Rating Score
first analgesic time | up to 24 hour after surgery
  the need of first analgesic after surgery
postoperative complications | up to 24 hour after surgery
  nausea-vomitting, motor block, hypertension, hypotension etc.
mobilization time | up to 24 hour after surgery
  when the patient is first mobilized

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No